CLINICAL TRIAL: NCT04543630
Title: Maxillary Sinus Floor Augmentation in Diabetic Patients With Particulated Autogenous Bone Graft Compared With Advanced Platelet-rich Fibrin. A Randomized Controlled Trial
Brief Title: Maxillary Sinus Floor Augmentation in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Simon Storgård Jensen, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20200009
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Jaw, Edentulous, Partially; Diabetes
Keywords: Implant Dentistry; Sinus floor augmentation; Autogenous bone; Platelet-rich fibrin; Diabetes
MeSH Terms: conditions — Jaw, Edentulous, Partially; Diabetes Mellitus | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Well-controlled diabetic patients with indication of sinus floor augmentation to allow placement of a dental implant in the posterior maxilla will be randomized to one of two sinus augmentation protocols: particulated autogenous bone or advanced platelet-rich fibrin
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to which arm the individual participant was treated under
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Particulated autogenous bone (Active Comparator): Particulated autogenous bone is considered the gold standard for sinus floor augmentation. The bone will be harvested locally
  Interventions: Procedure: Sinus floor augmentation
- Advanced platelet-rich fibrin (Experimental): Advanced platelet-rich fibrin will be be obtained through a blood sample from the participant
  Interventions: Procedure: Sinus floor augmentation

INTERVENTIONS:
Procedure: Sinus floor augmentation — Sinus floor augmentaion using the lateral window technique

SUMMARY:
Placement of implants in diabetic patients is associated with higher risk of implant failure and peri-implant marginal bone loss due to an increased susceptibility to infections, impaired wound healing and associated microvascular complications. However, diabetic patients do not encounter a higher implant failure rate compared with non-diabetic patients, if the plasma glucose levels are normal.

Prosthetic rehabilitation of the posterior maxilla with implants is frequently compromised due to atrophy of the alveolar process and pneumatisation of the maxillary sinus. Maxillary sinus floor augmentation (MSFA) with autogenous bone graft is generally considered the preferred grafting material due to its osteoinductive, osteogenic, and osteoconductive properties. However, harvesting of autogenous bone graft is associated with risk of donor site morbidity and unpredictable resorption of the graft. Thus, bone substitutes, blood coagulum and platelet rich fibrin are used increasingly to simplify the surgical procedure.

Fabrication of advanced platelet rich fibrin (APRF) from blood samples possess significant potential for bone regeneration without the use of additional autogenous bone grafts or bone substitutes. Consequently, use of APRF in conjunction with MSFA will avoid bone harvesting and simplify the surgical procedure.

The objective is to test the H0-hypothesis of no difference in implant treatment outcome after MSFA with particulated autogenous bone graft compared with APRF. Forty consecutively insulin-dependent diabetes patients with missing posterior maxillary tooth/teeth will be allocated to implant placement and MSFA with particulated autogenous bone graft from the zygomatic buttress or APRF. Blood samples will be obtained preoperatively and postoperatively. Clinical and radiographical evaluation using periapical radiographs and CBCT will be performed preoperatively, immediate postoperatively, before abutment connection, after prosthetic rehabilitation, one year, three years and five years after loading to assess the implant treatment outcome and the volumetric changes of the augmented area. Outcome measures will include survival of suprastructures and implants, volumetric stability of the augmented area, peri-implant marginal bone level, immunological analyses of blood samples, oral health related quality of life, and complications related to the two treatment modalities.

DETAILED DESCRIPTION:
Purpose The aim of the present study is to test the H0-hypotheisis of no difference in implant treatment outcome after MSFA in partial edentulous diabetic patients with particulated autogenous bone graft compared with APRF after five years of functional implant loading.

Objective

The objective is to test the H0 hypothesis of no differences in:

* Survival of suprastructures and implants.
* Volumetrical stability of the graft material.
* Peri-implant marginal bone level.
* Implantat stability quotient.
* Effect of implant placement and graft material on hematological and inflammatory parameters.
* Patient-reported outcome measures.
* Biologic and technical complications.

Outcome measures

* Survival of suprastructures. Loss of suprastructures is defined as a total loss because of a non-treatable mechanical/or biological complication.
* Survival of implants. Loss of implants is defined as removal of a non-integrated implant, mobility of previously clinical osseointegrated implant, and removal of non-mobile implants due to progressive peri-implant marginal bone loss and inflammation.
* Volumetric changes of the graft material.
* Peri-implant marginal bone level.
* Levels of hematological and inflammatory parameters.
* Patient-reported outcome measures.
* Biologic and technical complications e.g. loosening of crown and fractures of veneer ceramic.

Materials and methods Study population Forty consecutive insulin-dependent diabetes patients with missing posterior maxillary tooth/teeth will be included and randomly allocated to MSFA with particulated autogenous bone graft (control group) or APRF (test group). The study will be conducted at the Department of Odontology, Sections of Oral and Maxillofacial Surgery and Periodontology, University of Copenhagen and Department of Oral and Maxillofacial Surgery, Copenhagen University Hospital (Rigshospitalet) and Aalborg University Hospital, Aalborg, Denmark.

Ethical considerations, perspectives and informed consent The study has been approved by The North Denmark Region Committee on Health Research Ethics and will be performed according to the Declaration of Helsinki on clinical research. All patients will receive verbal and written information about the study by the investigators at a clinical visit prior to surgery. Written informed consent is mandatory for inclusion in the study and will be obtained by the investigators prior to surgery from each patient.

Initial examination

The initial examination of the patient will include:

* Clinical examination and assessment of the periodontal health status:
* Missing one posterior maxillary tooth (>4 months).
* Need of one implant in the posterior part of the maxilla.
* Adjacent tooth in opposite jaw in contact with planned crown.
* Plaque and gingival index, probing pocket depth, and probing attachment level of the adjacent tooth/teeth.
* Radiographical examination of the residual alveolar bone height based on CBCT.
* Orthopantomography to document the pre-treatment status.
* Blood samples.
* Patient will fill out the OHIP-14 questionnaire.

Surgical procedure The surgical procedure will be performed in local anesthesia with or without oral sedation or in general anesthesia. Implant installation and fabrication of the subsequently prosthetic solution will be performed according to manufacturer's recommendations. Prior to surgery, patients are pre-medicated as outlined in Table I. Patients will rinse with 0.12% chlorhexidine solution for one minute immediately before surgery. A sealed randomization envelope is opened in order to allocate patients to particulated autogenous bone graft from the zygomatic buttress (control) or APRF (test). Venous blood is collected from all the included patients via venipuncture of the forearm. The first 30 ml venous blood is discarded to prevent infection. A venous blood sample (80 ml, distributed in eight 10-ml glass-coated plastic tubes) via puncture of a vein in the cubital fossa is collected and centrifuged (A-PRF 12, Process, Nice, France) according to a previously described method. The blood samples are centrifuged at 200 g for 14 min. The tubes containing the centrifuged blood are placed to rest for approximately 25 min to give the fibrin clot a firmer consistency before collecting it for the final membrane preparation.

The maxillary sinus wall is exposed by an intraoral marginal incision from tuber maxillae to the first premolar with a vertical releasing incision. A 1 x 1 cm bony window to the maxillary sinus is created maintaining an intact Schneiderian membrane. The Schneiderian membrane is elevated from the sinus floor as well as the lateral sinus wall and displaced dorsocranially with blunt dissector. An implant bed is successively prepared on the top of the alveolar crest following manufactory's recommendations. An implant (AstraTech, 13 mm) is inserted with a cover screw. The implant stability quotient is measured for all inserted implants (Penguin, Integration Diagnostics Sweden AB, Göteborg, Sweden). Autogenous bone graft is harvested with curved SafeScraper from the zygomatic buttress. Specially prepared stainless steel cup are used to estimate 2 cm3 of particulated autogenous bone graft, which is packed around the inserted implant. In the test group, the sinus is filled with APRF membrane around the inserted implant. The bony window to the maxillary sinus is covered with a barrier membrane to seal the opening to the maxillary sinus. Periosteum and mucosa are sutured with a monofilament 4-0 suture. Minor perforations of sinus membrane will be covered with a membrane. If the sinus membrane is largely perforated, the procedure will be cancelled, and the patient will be withdrawn from the study. No provisional restoration is inserted during the healing period. Patients will be instructed to rinse with 0.12% chlorhexidine solution twice a day until suture removal has taken place after 7-10 days. Postoperative medication is outlined in Table I. Patient questionnaire will be filled out after one week and one month

Abutment surgery After six months of healing, abutment surgery is performed. The implant stability quotient is measured for all inserted implants. The implant is rinsed with saline and a prefabricated healing abutment is placed. The implants are manually tested for mobility and osseointegration by percussion. Mucosa is adapted and sutured with a monofilament 4-0 suture. The prosthetic restoration will be initiated three weeks after the healing abutment has been placed.

Prosthetic restoration Prosthetic restoration will include an individualized abutment and a fixed restoration performed by experienced prosthodontists with extensive clinical experience with implant-based prosthetics.

Clinical assessment

Patients will be scheduled for a postoperative clinical examination at baseline, one year, three year and five years after loading. The following parameters will be recorded at each visit:

* Plaque and gingival index, probing pocket depth, and probing attachment level.
* Oral health related quality of life - OHIP-14.
* Patient satisfaction (VAS).

Oral health related quality of life - OHIP-14 and patient satisfaction Oral Health Impact Profile (OHIP) is a questionnaire designed to measure impairment of oral health related quality of life and focuses on the frequency of complaints regarding the general dentition over a course of time. OHIP has been translated to and validated in several languages, including Danish. However, OHIP states the patient's overall oral impairment, and does not take a specific treatment site into account. Therefore, additional questionnaire including VAS may be used to evaluate the area of a missing tooth and/or a tooth replacement. The total implant treatment, peri-implant soft tissues, implant crown, and implant function at the follow-up examination will be assessed using a systematic questionnaire. Each question will be scored on a 100-mm VAS with 0 indicating extreme dissatisfaction and 100 indicating complete satisfaction. The VAS scores will be measured to the nearest mm by a ruler.

Hematological and inflammatory parameters The inflammatory assessment will include six blood samples obtained at inclusion, intraoperatively, one month postoperatively, at baseline, one year and five years after functional implant loading. Serum level of high sensitivity CRP (hsCRP9 (reference value 0-5 mg/L), fibrinogen (reference value 200-400 mg/dL), serum level of total cholesterol (standard ≤ 190 mg/dL), low-density lipoprotein (LDL-C) (standard ≤ 115 mg/dL), high-density lipoprotein (HDL-C) (standard for men > 40 mg/dL, for women > 46 mg/dL), leukotriene B4, prostaglandin E2, penetraxin-3, surfactant protein-D and serum levels of complement components C1, C3 and C9. White blood cell count (WBC) will be determined in blood from the heparin tube (standard 4.0-11.0 × 103 μL) following fractionation. Moreover, plasma levels of interleukin (IL)-1beta, IL-6, IL-10, tumor necrosis factor-alfa (TNF-alfa), transforming growth factor beta-1 (TGF-beta1), receptor activator of nuclear factor kappa-B ligand (RANKL) and osteoprotegrin (OPG), will be determined from plasma.

Radiographical assessment Radiographical evaluation will include seven sets of periapical radiographs and CBCT (I-Cat, Cone Beam 3-D Imaging System, Imaging Sciences, International Inc. Hatfield, USA) obtained preoperatively, immediately postoperatively, after abutment connection, at baseline, one year, three years and five years after loading. To provide blinding of the radiographical evaluation, the CBCT-scans are coded. Volumetrical changes of the grafts are estimated by point counting and the method described originally by Cavalieri. The original outline of the maxillary sinus before implant installation is recorded and superimposed on the corresponding images. A point grid test system is superimposed at random on all images, allowing 100-200 points to hit the graft of each maxillary sinus. The numbers of intersections over the graft are counted on each selected image. Cavalieri volume estimation principle is used to estimate the total volume of the graft.

Peri-implant marginal bone changes are evaluated by linear measurements on digital periapical radiographs and will be done on radiographs obtained at implant placement, baseline, 3-years and 5-years after loading. The distance from the implant-abutment connection to the marginal bone level will be measured mesially and distally parallel with the long-axis of the implant.

Data management and analysis, including calculation of sample size Data management and analysis including calculation of descriptive statistics are done using STATA (Data analysis and statistical software, version 13, StataCorp P, Texas, USA). A power calculation are based on differences in marginal bone level changes preformed in a previous study involving replacement of a single tooth with 2 different protocols of implant treatment.38 The calculation is based on the observed changes in marginal bone level from insertion of the implant to abutment connection (a change of 0.65 mm and a standard deviation of 0.65), 17 patients in each group reaches a power of 97% at the 5%-level. With 15% to cover drop-outs, each treatment group should include 20 patients. The statistical evaluation is performed by analysis of variance. Scheffe´s multiple comparison test is used post hoc to determine the relative effect of the various graft types. Level of significance is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years.
* Insulin-dependent diabetes with missing posterior maxillary tooth/teeth.
* Residual bone height of the maxillary alveolar process between 4 and 7 mm.
* Width of the alveolar process ≥6.5 mm.
* Presence of mandibular occluding teeth.
* Plasma glucose levels below 7.8 mmol/l or 140 mg/dl.

Exclusion Criteria:

* Contraindications to implant therapy.
* Full mouth plaque score >25%.
* Progressive periodontitis.
* Acute infection in the area intended for implant placement.
* Parafunction, bruxism, or clenching.
* Psychiatric problems or unrealistic expectations.
* Smoking. Previous smoker will not be excluded.
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 1 year
  Presence of implant at follow-up
Implant survival | 3 years
  Presence of implant at follow-up
Implant survival | 5 years
  Presence of implant at follow-up

SECONDARY OUTCOMES:
Volumetrical stability of the graft material | 1, 3 and 5 years
  Augmented volume measeured on CBCT
Peri-implant marginal bone level | 1, 3 and 5 years
  Marginal bone level measured on periapical radiographs
Effect of implant placement and graft material on hematological and inflammatory parameters | Pre-surgery, immediately after surgery, Baseline, 1, 3 and 5 years
  Inflammatory markers measuered through blood samples

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Dept. of Oral & Maxillofacial Surgery, Aalborg
  - Copenhagen University Hospital, Copenhagen
  - University of Copenhagen, School of Dental Medicine, Copenhagen

IPD SHARING:
Plan to Share IPD: No